CLINICAL TRIAL: NCT01938651
Title: Ultra-High Field (7 Tesla) MRI/MRS Evaluation of Breast Cancer
Brief Title: Ultra High Field MRI and MRS Techniques in Diagnosing Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding ceased
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Thomas Yankeelov, Director of Cancer Imaging Research, Vanderbilt University Institute of Imaging Science (VUIIS); Associate Professor of Radiology and Radiological Sciences, Biomedical Engineering, Physics and Astronomy, and Cancer Biology;, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VICC BRE 1277; NCI-2013-00435 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (7T ultra high-field MRI/MRS) (Experimental): Patients undergo measurement of tumor perfusion and permeability using DCE-MRI, tumor cellularity using DW-MRI, phospholipid metabolism using 31P MRS, macromolecular content using MT-MRI, and cellular protein content using CEST-MRI. All of these procedures are integrated into a single MRI exam lasting under 60 min.
  Interventions: Procedure: high field strength magnetic resonance imaging; Procedure: magnetic resonance spectroscopic imaging; Procedure: chemical exchange saturation transfer magnetic resonance imaging; Procedure: diffusion-weighted magnetic resonance imaging; Procedure: dynamic contrast-enhanced magnetic resonance imaging

INTERVENTIONS:
Procedure: high field strength magnetic resonance imaging — Undergo 7T MRI
  Other Names: high field strength MRI
Procedure: magnetic resonance spectroscopic imaging — Undergo 31P MRS
  Other Names: 1H-nuclear magnetic resonance spectroscopic imaging; Proton Magnetic Resonance Spectroscopic Imaging
Procedure: chemical exchange saturation transfer magnetic resonance imaging — Undergo CEST-MRI
  Other Names: CEST MRI
Procedure: diffusion-weighted magnetic resonance imaging — Undergo DW-MRI
  Other Names: diffusion-weighted MRI
Procedure: dynamic contrast-enhanced magnetic resonance imaging — Undergo DCE-MRI
  Other Names: DCE-MRI

SUMMARY:
This pilot clinical trial studies ultra-high field magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS) techniques in diagnosing breast cancer. New diagnostic procedures may be a more sensitive way to detect breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To implement quantitative dynamic contrast-enhanced (DCE)-MRI, diffusion-weighted (DW)-MRI, 31 phosphorus (31P) MRS, magnetization transfer (MT)-MRI, chemical exchange saturation transfer (CEST)-MRI, and high-resolution structural imaging at 7 Tesla in patients for diagnosing breast tumors.

OUTLINE:

Patients undergo measurement of tumor perfusion and permeability using DCE-MRI, tumor cellularity using DW-MRI, phospholipid metabolism using 31P MRS, macromolecular content using MT-MRI, and cellular protein content using CEST-MRI. Diagnostic performance of one, or a combination, of these metrics will be investigated in the context of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have signed an approved consent form
* Must be at least 18 years old
* Subjects must have undergone x-ray mammography and/or ultrasonography
* Subjects must have undergone standard clinical (1.5 Tesla) MRI as part of their standard-of-care diagnostic workup:

  * To evaluate the extent of disease for a previously diagnosed cancer, or
  * To evaluate a clinically suspected lesion that was occult on mammography and/or ultrasonography, or
  * Because the patient is considered high-risk (according to National Comprehensive Cancer Network [NCCN] criteria)
* Subjects must be classified Breast Imaging-Reporting and Data System (BI-RADS) 4 or 5
* Subjects must be scheduled for diagnostic biopsy to evaluate a lesion that measures >10 mm in the greatest dimension.

Exclusion Criteria:

* Subjects who have distant metastases
* Subjects who have any type of bioimplant activated by mechanical, electronic, or magnetic means (e.g., cochlear implants, pacemakers, neurostimulators, biostimulators, electronic infusion pumps, aneurysm clip, etc), because such devices may be displaced or malfunction
* Subjects who have any type of ferromagnetic bioimplant that could potentially be displaced by the magnetic field of the MRI scanner
* Subjects who may have shrapnel imbedded in their bodies (such as from war wounds), metal workers, and machinists (potential for metallic fragments in or near the eyes)
* Subjects with a history of renal disease (including renal cancer), diabetes, or human immunodeficiency virus (HIV)
* Creatinine >= 1.5 times upper limit of normal
* Estimated glomerular filtration rate < 30 mL/min
* Subjects who are pregnant or breast-feeding; the MRI Procedure Screening Form will be used to identify and exclude subjects who are pregnant or breastfeeding; a urine pregnancy test/or serum human chorionic gonadotropin (HCG) will also be performed for pre-menopausal women who are not using contraceptives
* Subjects who have exhibited past allergic or other adverse reactions in response to intravenous injection of Magnevist (gadopentetate dimeglumine) or other gadolinium-containing contrast agents
* Subjects who exhibit noticeable anxiety and/or claustrophobia or who exhibit severe vertigo when they are moved into the magnet bore
* Subjects incapable of giving informed written consent, for the following reasons:

  * Inability to adhere to the experimental protocols for any reason
  * Inability to communicate with the research team
  * Limited ability to give informed consent due to mental disability, altered mental status, confusion, or psychiatric disorders
  * Prisoners or other individuals deemed to be susceptible to coercion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity | At time of imaging procedure
  Ninety-percent simultaneous confidence rectangles for sensitivity and specificity will be constructed at the 25th, 50th (median), and 75th percentiles of the model predicted probability of disease.

SECONDARY OUTCOMES:
Pathological disease status | At time of imaging procedure
  A generalized linear mixed models analysis of variance with a logit link will be used to predict pathological disease status from MRI and MRS parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Yankeelov, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Related Info — http://www.vicc.org/ct/